CLINICAL TRIAL: NCT05853237
Title: Class iv Versus Class Iiib Laser Therapy on Median Sternotomy Healing After Coronary Artery Bypass Graft: a Randomize Control Trail
Brief Title: Class iv Versus Class Iiib Laser Therapy on Median Sternotomy Healing After Coronary Artery Bybass Graft
Acronym: wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidy F. Ahmed (Other)
Responsible Party: Sponsor-Investigator, Heidy F. Ahmed, physical therapy doctor wound care specialist at Al kasr Al Anini university hospital, Cairo , Egypt, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003308
Record Dates: First submitted 2023-04-06; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Wound; Wound Heal; Wound Infection
Keywords: Coronary arteries bypass grafting; high level laser therapy; Low-level laser therapy; Median sternotomy healing
MeSH Terms: conditions — Wounds and Injuries; Wound Infection | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: group A receive laser therapy class IV+traditional wound care and group (B): Laser therapy class IIIb + traditional wound care and group C receive only traditional wound care
Who Masked: Participant, Outcomes Assessor
Masking Description: he patientsdidnt know the different types of laser which procedure they received & the outcomes assessor done by my supervisors and didn't know which result related to specific group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- class IV group (Experimental): start from day one surgery for 4 successive weeks, the goal in the phase I (1st 10 days after surgery) is decontamination, improve circulation, pain reduction &wound healing acceleration The goal of phase II (next10 days till complete healing) is improve osteo-integration, pain reduction & enhance superficial collagen production to decrease scarring. The parameters are: Power > 500 mW; fluence 20 joule/ cm2 with (980, 915, 810 nm) and 5 joules/ cm2 by 650 nm; mode (continuous); hand piece radius = 2.5 cm; spot size (Area) = 5 cm; application by scanning not spotting to avoid thermal effect and time of session is 5- 10 minutes
  Interventions: Device: laser therapy for wound management
- class IIIb (Experimental): Use the same protocol as in HLLT with the same wave lengths but with low power Power = 200- 300 mW; fluence 20 joule/ cm2 with (980, 915, 810 nm) and 5 joules/ cm2 by 650 nm; mode (continuous); hand piece radius = 2.5 cm; spot size (Area) = 5 cm; application by spotting and time of session was 25- 30 minutes.
  Interventions: Device: laser therapy for wound management
- traditional wound care (Active Comparator): According to the hospital protocol Irrigation of the wound by normal saline, betadine application, bivatracin spray and Change dressing daily to protect the wound from infection
  Interventions: Device: laser therapy for wound management

INTERVENTIONS:
Device: laser therapy for wound management — comparison between laser effect on post median sternotomy incision compared to traditional wound care

SUMMARY:
LASER therapy is potent physiotherapy modalities, providing better sternotomy healing for patients who have undergone CABG surgery, compared with traditional wound care management alone. HLLT and LLLT were found to be the most effective methods for sternotomy healing post-CABG surgery, with HLLT offering superior performance in the case of the high deep penetration and significance less time needed to deliver the same joules/ cm compared to LLLT used for the wound site.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of class IV high-level laser therapy (HLLT) versus class IIIb low level laser therapy (LLLT) on sternotomy healing following coronary artery bypass grafting (CABG) surgery. Forty- five patients male patients who had CABG surgery in the age range of 45-65 years were divided randomly into three equal groups (n = 15). The group HLLT laser received HLLT plus traditional wound management, while the group LLLT laser received LLLT plus traditional wound management. The control group only received a traditional wound management in form of saline irrigation, dressing, and topical bivatracin spray according to hospital protocol. All groups were offered 10 sessions over 4 weeks. HLLT and LLLT were found to be the most effective methods for sternotomy healing post-CABG surgery, with HLLT offering superior performance in the case of the high deep penetration and significance less time needed to deliver the same joules/ cm compared to LLLT used for the wound site.

ELIGIBILITY:
Inclusion Criteria:

* aged between 45 and 65 years
* male gender; haemodynamic stability
* body mass index (BMI) from 18.5 to 29.9 kg/m2
* Non-infected sternotomy site
* Normal ejection fraction to ensure normal vascularity.

Exclusion Criteria:

* included previous thoracic surgery
* emergency or urgent coronary artery bypass surgery
* respiratory insufficiency after surgery, manifesting hypoxemia with partial oxygen pressure in arterial blood < 60 mmHg; Ejection fraction < 50%
* Paramedian sternotomy which may cut wire causing sternal mobilization which is the start of deep wound infection
* Bilateral mammary harvesting which decrease blood flow to sternum; low cardiac output syndrome with ST segment elevation in multiple electrocardiogram leads, cardiac arrhythmias or hypotension, according to the American College of Cardiology Foundation and American Heart Association
* other medical conditions, such as diabetes, uncontrolled hypertension and obesity.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all the inclusion criteria are male patients
Enrollment: 45 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
PUSH pressure ulcer scaling healing score for wound healing | two consecutive months
  measure wound surface area in cm 2
PUSH pressure ulcer scaling healing score for wound healing | two consecutive months
  measure wound exudate in percent

SECONDARY OUTCOMES:
VAS visual analogue scale | two consecutive months
  visual analogue scale of the pain in numbers from 1-10(10 max pain and 1 min pain)

CONTACTS AND LOCATIONS:
Overall Officials: Heidy F Ahmed, master, Principal Investigator — Kasr al aini
Locations (1):
- Kasr Al Aini University Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD), all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: In the next month of registration.
Access Criteria: Information will be available upon request through the following e-mail: heidy.fouad@gmail.com.

REFERENCES:
- [Background] Sanchis-Gomar F, Perez-Quilis C, Leischik R, Lucia A. Epidemiology of coronary heart disease and acute coronary syndrome. Ann Transl Med. 2016 Jul;4(13):256. doi: 10.21037/atm.2016.06.33. PMID 27500157
- [Background] Olbrecht VA, Barreiro CJ, Bonde PN, Williams JA, Baumgartner WA, Gott VL, Conte JV. Clinical outcomes of noninfectious sternal dehiscence after median sternotomy. Ann Thorac Surg. 2006 Sep;82(3):902-7. doi: 10.1016/j.athoracsur.2006.04.058. PMID 16928505
- [Background] Cove ME, Spelman DW, MacLaren G. Infectious complications of cardiac surgery: a clinical review. J Cardiothorac Vasc Anesth. 2012 Dec;26(6):1094-100. doi: 10.1053/j.jvca.2012.04.021. Epub 2012 Jul 4. No abstract available. PMID 22765993
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825
- [Background] Brocki BC, Thorup CB, Andreasen JJ. Precautions related to midline sternotomy in cardiac surgery: a review of mechanical stress factors leading to sternal complications. Eur J Cardiovasc Nurs. 2010 Jun;9(2):77-84. doi: 10.1016/j.ejcnurse.2009.11.009. Epub 2010 Jan 3. PMID 20051323
- [Background] Chang VT, Sorger B, Rosenfeld KE, Lorenz KA, Bailey AF, Bui T, Weinberger L, Montagnini M. Pain and palliative medicine. J Rehabil Res Dev. 2007;44(2):279-94. doi: 10.1682/jrrd.2006.06.0067. PMID 17551879
- [Background] Amaroli A, Ravera S, Baldini F, Benedicenti S, Panfoli I, Vergani L. Photobiomodulation with 808-nm diode laser light promotes wound healing of human endothelial cells through increased reactive oxygen species production stimulating mitochondrial oxidative phosphorylation. Lasers Med Sci. 2019 Apr;34(3):495-504. doi: 10.1007/s10103-018-2623-5. Epub 2018 Aug 25. PMID 30145725
- [Background] 9. Pryor BA. Advances in Laser Therapy for the treatment of work related injuries. Current Perspectives in Clinical Treatment and Management onWorkers' Compensation Cases, 1st edn. Bentham Science Publishers Ltd. 2011 Apr 23:191-201.
- [Background] Liao X, Xie GH, Liu HW, Cheng B, Li SH, Xie S, Xiao LL, Fu XB. Helium-neon laser irradiation promotes the proliferation and migration of human epidermal stem cells in vitro: proposed mechanism for enhanced wound re-epithelialization. Photomed Laser Surg. 2014 Apr;32(4):219-25. doi: 10.1089/pho.2013.3667. Epub 2014 Mar 24. PMID 24661127
- [Background] Veith AP, Henderson K, Spencer A, Sligar AD, Baker AB. Therapeutic strategies for enhancing angiogenesis in wound healing. Adv Drug Deliv Rev. 2019 Jun;146:97-125. doi: 10.1016/j.addr.2018.09.010. Epub 2018 Sep 26. PMID 30267742
- [Background] 12. Johnson JF. Laser therapy and pain management. Laser Therapy in Veterinary Medicine: Photobiomodulation. 2017 May 11:75-87.
- [Background] Tucker LD, Lu Y, Dong Y, Yang L, Li Y, Zhao N, Zhang Q. Photobiomodulation Therapy Attenuates Hypoxic-Ischemic Injury in a Neonatal Rat Model. J Mol Neurosci. 2018 Aug;65(4):514-526. doi: 10.1007/s12031-018-1121-3. Epub 2018 Jul 22. PMID 30032397
- [Background] 14. Pryor BA. Advances in Laser Therapy for the treatment of work related injuries. Current Perspectives in Clinical Treatment and Management onWorkers' Compensation Cases, 1st edn. Bentham Science Publishers Ltd. 2011 Apr 23:191-201.
- [Background] Alayat MS, El-Sodany AM, Ebid AA, Shousha TM, Abdelgalil AA, Alhasan H, Alshehri MA. Efficacy of high intensity laser therapy in the management of foot ulcers: a systematic review. J Phys Ther Sci. 2018 Oct;30(10):1341-1345. doi: 10.1589/jpts.30.1341. Epub 2018 Oct 12. PMID 30349176
- [Background] 16. Mikołajczyk, Z., Nowak, I., Kawiński, A., & Mik, M. (2021). Phototherapy in the Treatment of Diabetic Foot-A Preliminary Study. Autex Research Journal, 21(4), 482-490.
- [Background] Fernandes GA, Lima AC, Gonzaga IC, de Barros Araujo R Jr, de Oliveira RA, Nicolau RA. Low-intensity laser (660 nm) on sternotomy healing in patients who underwent coronary artery bypass graft: a randomized, double-blind study. Lasers Med Sci. 2016 Dec;31(9):1907-1913. doi: 10.1007/s10103-016-2069-6. Epub 2016 Sep 20. PMID 27649961
- [Background] Coulson SE, Adams RD, O'Dwyer NJ, Croxson GR. Physiotherapy rehabilitation of the smile after long-term facial nerve palsy using video self-modeling and implementation intentions. Otolaryngol Head Neck Surg. 2006 Jan;134(1):48-55. doi: 10.1016/j.otohns.2005.09.010. PMID 16399180
- [Background] Hillis LD, Smith PK, Anderson JL, Bittl JA, Bridges CR, Byrne JG, Cigarroa JE, Disesa VJ, Hiratzka LF, Hutter AM Jr, Jessen ME, Keeley EC, Lahey SJ, Lange RA, London MJ, Mack MJ, Patel MR, Puskas JD, Sabik JF, Selnes O, Shahian DM, Trost JC, Winniford MD. 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Dec 6;124(23):2610-42. doi: 10.1161/CIR.0b013e31823b5fee. Epub 2011 Nov 7. No abstract available. PMID 22064600
- [Background] Hon J, Lagden K, McLaren AM, O'Sullivan D, Orr L, Houghton PE, Woodbury MG. A prospective, multicenter study to validate use of the PUSH in patients with diabetic, venous, and pressure ulcers. Ostomy Wound Manage. 2010 Feb 1;56(2):26-36. PMID 20200443
- [Background] El-Ansary D, Waddington G, Adams R. Trunk stabilisation exercises reduce sternal separation in chronic sternal instability after cardiac surgery: a randomised cross-over trial. Aust J Physiother. 2007;53(4):255-60. doi: 10.1016/s0004-9514(07)70006-5. PMID 18047460
- [Background] Sa MP, Silva DO, Lima EN, Lima Rde C, Silva FP, Rueda FG, Escobar RR, Cavalcanti PE. Postoperative mediastinitis in cardiovascular surgery postoperation. Analysis of 1038 consecutive surgeries. Rev Bras Cir Cardiovasc. 2010 Jan-Mar;25(1):19-24. PMID 20563463
- [Background] 23. Peplow P, Chung T, Baxter D. Application of low level laser technologies for pain relief and wound healing: Overview of scientific bases. Phys Ther Rev. 2000;15:4.
- [Background] Bashardoust Tajali S, Macdermid JC, Houghton P, Grewal R. Effects of low power laser irradiation on bone healing in animals: a meta-analysis. J Orthop Surg Res. 2010 Jan 4;5:1. doi: 10.1186/1749-799X-5-1. PMID 20047683
- [Background] Helmy ZM, Mehani SHM, El-Refaey BH, Al-Salam EHA, Felaya EEE. Low-level laser therapy versus trunk stabilization exercises on sternotomy healing after coronary artery bypass grafting: a randomized clinical trial. Lasers Med Sci. 2019 Aug;34(6):1115-1124. doi: 10.1007/s10103-018-02701-4. Epub 2018 Dec 13. PMID 30547261
- [Background] Kazemi Khoo N, Babazadeh K, Lajevardi M, Dabaghian FH, Mostafavi E. Application of Low-Level Laser Therapy Following Coronary Artery Bypass Grafting (CABG) Surgery. J Lasers Med Sci. 2014 Spring;5(2):86-91. PMID 25653805
- [Background] Renno AC, McDonnell PA, Parizotto NA, Laakso EL. The effects of laser irradiation on osteoblast and osteosarcoma cell proliferation and differentiation in vitro. Photomed Laser Surg. 2007 Aug;25(4):275-80. doi: 10.1089/pho.2007.2055. PMID 17803384
- [Background] 28. Baptista IDC, Chavantes MC, Dallan LDO, Stolf NAG (2009) Laser de baixa intensidade: nova tecnologia para os enfermeiros na cicatrizaçao pós-esternotomia. Rev Soc Cardiol Estado São Paulo 19:3-8
- [Background] Dixit S, Maiya A, Umakanth S, Borkar S. Photobiomodulation of surgical wound dehiscence in a diabetic individual by low-level laser therapy following median sternotomy. Indian J Palliat Care. 2013 Jan;19(1):71-5. doi: 10.4103/0973-1075.110242. PMID 23766600